CLINICAL TRIAL: NCT02903004
Title: Randomized Phase III Trial on Trabectedin (ET-743) vs Clinician's Choice Chemotherapy in Recurrent Ovarian, Primary Peritoneal or Fallopian Tube Cancers of BRCA Mutated or BRCAness Phenotype Patients
Brief Title: Trial on Trabectedin (ET-743) vs Clinician's Choice Chemotherapy in Recurrent Ovarian, Primary Peritoneal or Fallopian Tube Cancers of BRCA Mutated or BRCAness Phenotype Patients
Acronym: MITO23
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 986
Record Dates: First submitted 2016-08-26; First posted 2016-09-16 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Trabectedin; liposomal doxorubicin; Topotecan; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trabectedin (Experimental): Trabectedin 1.3 mg/m2 d1 q 21 in 3 hours (central line)
  Interventions: Drug: Trabectedin
- Standard Treatment (Other): Pegylated Liposomal Doxorubicin 40 mg/mq q 28 or Topotecan 4 mg/ m2 dd 1,8,15 q 28 or Gemcitabine 1000 mg/mq dd 1, 8, 15 q 28 Weekly Paclitaxel 80 mg/ m2 dd 1, 8, 15 q 28 Carboplatin AUC 5-6 q 21 or 28
  Interventions: Drug: Pegylated Liposomal Doxorubicin; Drug: Topotecan; Drug: Gemcitabine; Drug: Weekly Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Trabectedin
  Other Names: Yondelis
  Arms: Trabectedin
Drug: Pegylated Liposomal Doxorubicin
  Arms: Standard Treatment
Drug: Topotecan
  Arms: Standard Treatment
Drug: Gemcitabine
  Arms: Standard Treatment
Drug: Weekly Paclitaxel
  Arms: Standard Treatment
Drug: Carboplatin
  Arms: Standard Treatment

SUMMARY:
This is an open-label, prospective, multicenter, randomized Phase III, clinical trial evaluating the efficacy and safety of trabectedin in BRCA1 and BRCA2 mutation carrier and BRCAness phenotype advanced ovarian cancer patients in comparison to physician' choice chemotherapy.

Arm A: Trabectedin 1.3 mg/mq d1 q 21 in 3 hours (central line) Arm B: Pegylated Liposomal Doxorubicin 40 mg/mq q 28 or Topotecan 4 mg/mq dd 1,8,15 q 28 or Gemcitabine 1000 mg/mq dd 1, 8, 15 q 28 Weekly Paclitaxel 80 mg/mq gg 1, 8, 15 q 28 Carboplatin AUC 5-6 q 21 or 28

Patients will be randomly assigned in a 1:1 ratio to treatment arms. During the randomization process, patients will be stratified by

* Platinum sensitivity
* Measurable disease
* Number of previous chemotherapy lines > vs < 3
* BRCA mutational status

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio to receive one of the following treatments: Arm A: Trabectedin 1.3 mg/m2 d1 q 21 in 3 hours (central line) Arm B: Pegylated Liposomal Doxorubicin 40 mg/mq q 28 or Topotecan 4 mg/ m2 dd 1,8,15 q 28 or Gemcitabine 1000 mg/mq dd 1, 8, 15 q 28 Weekly Paclitaxel 80 mg/ m2 dd 1, 8, 15 q 28 Carboplatin AUC 5-6 q 21 or 28 Randomization will be stratified based on platinum-free interval (PFI) (PFI ≥ 0 and ≤ 6 months vs. PFI > 6 months), presence / absence of measurable disease/number of previous chemotherapy lines, germline BRCA mutational status vs BRCAness phenotype.

Platinum-free interval (PFI) is defined as the time from the last dose of the platinum containing regimen until the first date progression.

Subjects will continue to receive chemotherapy treatment until disease progression (clinical progression meant as global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression is considered progression of disease), intolerability, patient refusal, investigator decision or death from any cause.

Subjects will be evaluated every 12 weeks ± 1 week by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for objective radiographic response and radiographic disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Female of age 18 years or older
2. Histologically or cytologically documented invasive epithelial ovarian cancer, primary peritoneal carcinoma, or fallopian tube cancer
3. Platinum resistant or sensitive patients with either:

   1. BRCA mutated patients
   2. BRCAness phenotype patients: patients who have received and responded (subsequent PFI>6 months) to at least 2 previous platinum based chemotherapy lines
   3. Platinum sensitive patients who are not able to receive or not willing to receive other platinum treatments
4. Measurable and evaluable disease per RECIST 1.1(Subjects with isolated rising CA-125 without radiologically visible disease are excluded)
5. ECOG performance status 0 or 1
6. No limits in the number of previous chemotherapy lines, previous treatment with parp inhibitors is allowed
7. Left Ventricular Ejection Fraction (LVEF) ≥ institutional lower limit normal
8. Life expectancy of at least 3 months
9. Adequate organ functions:

   1. Hematopoietic: Absolute neutrophil count ≥ 1,500/mm3; Platelet count ≥ 100,000/mm3; Hemoglobin ≥ 9 g/dl
   2. Hepatic: AST and ALT ≤ 1.5 times upper limit of normal (ULN)* ; Alkaline Phosphatase ≤ 2.5 times ULN* ; Bilirubin ≤ 1.5 times ULN. NOTE: * ≤ 3 times ULN if liver metastases are present
   3. Renal: Creatinine Clearance ≥ 45 ml/min or Serum Creatinine ≤1.5 x ULN
   4. Serum Albumin >2.5 g/dl
10. No other invasive malignancy within the past 3 years except non-melanoma skin cancer or in situ cervical cancer (patients with previous cancers may be enrolled providing that no recurrences have be reported in the last 3 years)
11. Written Informed Consent
12. Adequately recovered from the acute toxicity of any prior treatment
13. For agents in the standard arm, also refer to the local prescribing information with regards to warnings, precautions, and contraindications

Exclusion Criteria:

1. Prior exposure to trabectedin
2. Known hypersensitivity to any of the components of the trabectedin i.v. formulation or dexamethasone
3. Subjects with borderline ovarian cancer, ie. Subject with low malignant potential tumors are excluded
4. Less than 2 reported responses to platinum (i.e. subsequent recurrences at least 6 months after the first and the second platinum based treatment), unless BRCA mutation is documented.
5. Less than 4 weeks from last dose of therapy with any investigational agent, or chemotherapy
6. History of another neoplastic disease (except basal cell carcinoma or cervical carcinoma in situ adequately treated) unless in remission for 3 years or longer
7. Known clinically relevant CNS metastases, unless treated and asymptomatic
8. Other serious illnesses, such as:

   1. Congestive heart failure or angina pectoris; myocardial infarction within 1 year before enrolment; uncontrolled arterial hypertension or arrhythmias.
   2. Psychiatric disorder that prevents compliance with protocol.
   3. Active viral hepatitis; or chronic liver disease.
   4. Active infection.
   5. Any other unstable medical conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 4 years
  The primary objective is to compare the Trabectedin versus physician' choice chemotherapy in terms of overall survival (OS).

SECONDARY OUTCOMES:
Progression free survival (PFS) | 4 years
  Progression-free survival [the diagnosis of progression will be assessed by radiological criteria; CA 125 increases alone (GCIG criteria of progression) will not be considered as progression of disease without a radiological confirmation of progression].
Duration of Response | 4 years
  Duration of response
Adverse events | 4 years
  Incidence of adverse events, according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Domenica Lorusso, Prof., Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Domenica Lorusso, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salutari V, Ferrandina G, Vincenzi B et al. Efficacy and safety outcomes in heavily pretreated patients (pts) with relapsed ovarian cancer (roc ) after single agent trabectedin. ASCO 2013, submitted.
- [Background] Monk BJ, Herzog T, Kay S et al. A randomized Phase III study of trabectedin with pegylated liposomal doxorubicin (PLD) versus PLD in relapsed, recurrent ovarian cancer (OC). Ann. Oncol. 19(Suppl. 8), (2009)
- [Background] K. L. Tedesco, J. L. Blum, A. Goncalves, J. Lubinski, N. Ben-Baruch, C. R. Osborne, P. Lardelli, A et al. phase II trial of trabectedin (T) in patients (pts) with HER2-positive and BRCA1/2 germ-line-mutated metastatic breast cancer (MBC). J Clin Oncol 28:15s, 2010 (suppl; abstr 1038)
- [Result] Takebayashi Y, Pourquier P, Zimonjic DB, Nakayama K, Emmert S, Ueda T, Urasaki Y, Kanzaki A, Akiyama SI, Popescu N, Kraemer KH, Pommier Y. Antiproliferative activity of ecteinascidin 743 is dependent upon transcription-coupled nucleotide-excision repair. Nat Med. 2001 Aug;7(8):961-6. doi: 10.1038/91008. PMID 11479630
- [Result] Damia G, Silvestri S, Carrassa L, Filiberti L, Faircloth GT, Liberi G, Foiani M, D'Incalci M. Unique pattern of ET-743 activity in different cellular systems with defined deficiencies in DNA-repair pathways. Int J Cancer. 2001 May 15;92(4):583-8. doi: 10.1002/ijc.1221. PMID 11304695
- [Result] Schoffski P, Taron M, Jimeno J, Grosso F, Sanfilipio R, Casali PG, Le Cesne A, Jones RL, Blay JY, Poveda A, Maki RG, Nieto A, Tercero JC, Rosell R. Predictive impact of DNA repair functionality on clinical outcome of advanced sarcoma patients treated with trabectedin: a retrospective multicentric study. Eur J Cancer. 2011 May;47(7):1006-12. doi: 10.1016/j.ejca.2011.01.016. Epub 2011 Mar 4. PMID 21376569
- [Result] Germano G, Frapolli R, Belgiovine C, Anselmo A, Pesce S, Liguori M, Erba E, Uboldi S, Zucchetti M, Pasqualini F, Nebuloni M, van Rooijen N, Mortarini R, Beltrame L, Marchini S, Fuso Nerini I, Sanfilippo R, Casali PG, Pilotti S, Galmarini CM, Anichini A, Mantovani A, D'Incalci M, Allavena P. Role of macrophage targeting in the antitumor activity of trabectedin. Cancer Cell. 2013 Feb 11;23(2):249-62. doi: 10.1016/j.ccr.2013.01.008. PMID 23410977
- [Result] del Campo JM, Sessa C, Krasner CN, Vermorken JB, Colombo N, Kaye S, Gore M, Zintl P, Gomez J, Parekh T, Park YC, McMeekin S. Trabectedin as single agent in relapsed advanced ovarian cancer: results from a retrospective pooled analysis of three phase II trials. Med Oncol. 2013 Mar;30(1):435. doi: 10.1007/s12032-012-0435-1. Epub 2013 Feb 9. PMID 23397080
- [Result] Erba E, Bergamaschi D, Bassano L, Damia G, Ronzoni S, Faircloth GT, D'Incalci M. Ecteinascidin-743 (ET-743), a natural marine compound, with a unique mechanism of action. Eur J Cancer. 2001 Jan;37(1):97-105. doi: 10.1016/s0959-8049(00)00357-9. PMID 11165136
- [Result] Herrero AB, Martin-Castellanos C, Marco E, Gago F, Moreno S. Cross-talk between nucleotide excision and homologous recombination DNA repair pathways in the mechanism of action of antitumor trabectedin. Cancer Res. 2006 Aug 15;66(16):8155-62. doi: 10.1158/0008-5472.CAN-06-0179. PMID 16912194
- [Result] Safra T, Borgato L, Nicoletto MO, Rolnitzky L, Pelles-Avraham S, Geva R, Donach ME, Curtin J, Novetsky A, Grenader T, Lai WC, Gabizon A, Boyd L, Muggia F. BRCA mutation status and determinant of outcome in women with recurrent epithelial ovarian cancer treated with pegylated liposomal doxorubicin. Mol Cancer Ther. 2011 Oct;10(10):2000-7. doi: 10.1158/1535-7163.MCT-11-0272. Epub 2011 Aug 11. PMID 21835933
- [Result] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Derived] Lorusso D, Raspagliesi F, Ronzulli D, Valabrega G, Colombo N, Pisano C, Cassani C, Tognon G, Tamberi S, Mangili G, Mammoliti S, De Giorgi U, Greco F, Mosconi AM, Breda E, Artioli G, Andreetta C, Casanova C, Ceccherini R, Frassoldati A, Salutari V, Giolitto S, Scambia G. Single-Agent Trabectedin Versus Physician's Choice Chemotherapy in Patients With Recurrent Ovarian Cancer With BRCA-Mutated and/or BRCAness Phenotype: A Randomized Phase III Trial. J Clin Oncol. 2024 May 1;42(13):1488-1498. doi: 10.1200/JCO.23.01225. Epub 2024 Feb 5. PMID 38315944